CLINICAL TRIAL: NCT06042868
Title: Effect of Implementing Emergency Nursing Protocol About Obstructive Anuria and Oliguria on Critically Ill Patients' Outcomes
Brief Title: Effect of Implementing Emergency Nursing Protocol About Oliguria and Anuria on Patients' Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hager AbdelNasser Hussein (Other)
Responsible Party: Sponsor-Investigator, Hager AbdelNasser Hussein, Mrs, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Oliguria and anuria managment
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Oliguria
MeSH Terms: conditions — Oliguria | interventions — Nursing Assessment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Nursing protocol — Emergency nursing protocol

SUMMARY:
This study is aim to evaluate the effect of implementing emergency nursing protocol of obstructive anuria and oliguria on critically ill patients' outcomes.

DETAILED DESCRIPTION:
Obstructive anuria is defined as a total cessation of diuresis or a volume of less than 200 ml /24 hours or 0 mL/12 h. Oliguria is defined as a urine output that is less than 400 mL/24 h or less than 17 mL/h, due to unilateral or bilateral blockage of a single anatomical or functional kidney. It is rapidly the cause of acute renal failure, endangering the vital prognosis in the short term and requiring emergency treatment in a specialized environment, whatever its etiology (Afifi R, et al., 2022).

Obstructive anuria and oliguria constitutes a major cause for surgical acute kidney injury (AKI) due to several diseases as cervical cancer, urinary stone, bladder cancer, urinary tract stenosis, and iatrogenic causes. However, Obstructive anuria and oliguria management varies between each case; the treatment of choice is based on each patient's condition. We discovered that a proper management of obstructive anuria resulted in a low mortality rate as well as restoration of renal function in most patients (Wicaksono F, et al., 2021).

Anuria /Oliguria is frequently observed in the perioperative period and may be the consequence of hypovolemia and/or pain, both triggering the sympathetic nervous system, which in turn lead to activation of the renin-angiotensin-aldosterone system with ensuing oliguria. However, oliguria may also represent a warning of deteriorating renal function, especially in critically ill patients (Vincent JL and et al., 2020).

2

There are many complications from anuria and oliguria as cardiovascular complications include congestive heart failure, pulmonary edema, and hypertension, mainly as a result of salt and water retention. Gastrointestinal complications as anorexia, nausea, vomiting and gastrointestinal bleeding. Neurologic complications as confusion and seizures may develop in the course of acute oliguria. Impaired defenses and responses against infection due to uremia and inappropriate use of antibiotics may contribute to the high degree of infectious complications. Percutaneous nephrostomy is an excellent initial procedure to relieve obstruction with minimal complications. The second choice is renal dialysis for deteriorated patients (Rachid M, et al., 2020).

There is a critical role of nurse for taking history for oliguria and anuria as total volumes of urine in 24 h, color of urine, accompanying symptoms as (frequency, urgency and dysuria), special food or drugs as (nephrotoxic drugs, chemicals, eating raw fish guts); history of relevant diseases as (hemorrhoea, shock, heart failure, renal percussive pain, high fever, etc.) ; Past history including respiratory infection, angina, chronic nephritis, urinary calculus, prostate hyperplasia; travelling history as (epidemic hemorrhagic fever or epidemic area) should be pay attention. Critical care nurse must monitor hemodynamic parameters, signs of dehydration or fluid overload, fluids balances and duration of oliguria

ELIGIBILITY:
Inclusion Criteria Diagnosis: Post renal oliguria and anuria for 12 hours. Investigations: serum creatinine < 2 mg. Exclusion Criteria Patients who refused participation in study. Patients who drained by PCN. Patients who dialysate > 1 session. Patients with GCS <12

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Complications | 1year
  Electrolytes disturbances and renal failure